CLINICAL TRIAL: NCT06478719
Title: A Phase I/II Randomized, Double-blinded Study of FB-1603 to Evaluate the Safety and Efficacy in Hepatocellular Carcinoma Patients Receiving Transarterial Chemoembolization (FECHT Trial)
Brief Title: To Evaluate Safety and Efficacy of FB-1603 in Hepatocellular Carcinoma Patient Receiving Transarterial Chemoembolization
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Febico Biomedical Corp. (Industry)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: FB-1603_TACE_PII_2022_1
Record Dates: First submitted 2024-06-17; First posted 2024-06-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- placebo (Placebo Comparator): 4*Placebo oral capsule each time, TID (three times a Day). treatment period: start two weeks before TACE until eight weeks after TACE.
  Interventions: Drug: Placebo
- low dose FB-1603 (990mg/day) (Experimental): 2*FB-1603 165 mg oral capsule and 2*Placebo oral capsule each time, TID (990 mg/day). treatment period: start two weeks before TACE until eight weeks after TACE.
  Interventions: Drug: Placebo; Drug: FB-1603
- high dose FB-1603 (1980mg/day) (Experimental): 4*FB-1603 165 mg oral capsule each time, TID (1980 mg/day). treatment period: start two weeks before TACE until eight weeks after TACE.
  Interventions: Drug: FB-1603

INTERVENTIONS:
Drug: Placebo — Placebo oral capsule
  Arms: low dose FB-1603 (990mg/day); placebo
Drug: FB-1603 — FB-1603 (165 mg/cap) oral capsule
  Arms: high dose FB-1603 (1980mg/day); low dose FB-1603 (990mg/day)

SUMMARY:
The goal of this clinical trial is to assess the efficacy of FB-1603 on improving liver function impairment in hepatocellular carcinoma patients receiving transarterial chemoembolization. The main question it aims to answer is:

Changes in the level of liver function parameters, including AST, ALT, or total bilirubin, from baseline to Visit 3, Visit 4, Visit 5, and Visit 6

There is a comparison group: Researchers will compare arm 1 placebo to see if FB-1603 is work to treat the liver function.

Participants will

1. Take drug FB-1603 990mg/day, FB-1603 1980mg/day or a placebo every day for 10 weeks.
2. Visit the clinic on day 4, 7, 10, 14, 28, 56 and 84 (follow-up)

DETAILED DESCRIPTION:
I. Objectives:

* Primary objective: To assess the efficacy of FB-1603 on improving liver function impairment after transarterial chemoembolization (TACE) in subjects
* Secondary objective:

  * To evaluate the safety of FB-1603 in subjects
  * To evaluate selected parameters indicative of clinical efficacy
  * To assess postembolization syndrome improvement of FB-1603 compared with placebo
  * To evaluate virologic test level of FB-1603 compared with placebo
  * To assess liver stiffness change of FB-1603 compared with placebo
* Exploratory objective:

  * To assess the antioxidation activity of FB-1603 in hepatocellular carcinoma (HCC) subjects after TACE

II. Investigational product:

1. Name: FB-1603 oral capsule (FB-1603)
2. Dosage form: 165 mg oral capsule
3. Dose(s): Each arm consisted of 40 subjects.

   * Arm 1: 4*Placebo each time, TID (three times a Day), two weeks before and eight weeks after TACE
   * Arm 2: 2*FB-1603 165 mg oral capsule and 2*Placebo each time, TID (990 mg/day), two weeks before and eight weeks after TACE
   * Arm 3: 4*FB-1603 165 mg oral capsule each time, TID (1980 mg/day), two weeks before and eight weeks after TACE
4. Dosing schedule:

   All enrolled subjects will be randomly assigned (1:1:1) to receive low dose (990 mg/day), high dose (1980 mg/day) of FB-1603 165 mg oral capsule or placebo capsule three times a day for 10 weeks. Each subject starts receiving FB-1603 165 mg oral capsule or placebo capsule on two weeks before and eight weeks after TACE. The investigational drugs should be taken orally about 10 minutes before the breakfast, lunch, and dinner
5. Mechanism of action:

The proposed mechanism is that FB-1603 can improve liver function via decrease of oxidative stress. In previous study conducted in diethylnitrosamine (DEN) induced liver cirrhosis and cancer rat model (Report #: FENTU30SEP2009) shown that the extent of oxidative stress determined by NBT (Nitro blue tetrazolium) staining was significant decreased in treatment group orally administrated with 0.8, 1 or 2 g/kg/day of FB-1603 compared with the control group.

III. Developmental phase: phase I and II

IV. Study design:

1. placebo control study
2. Blinding: double blind
3. Randomized: yes
4. Parallel
5. Duration of treatment: days 10 weeks months years
6. Titration: forced
7. Single center

VI. Study procedures:

This is a randomized, double-blind, 10-week dose-finding study in 3 parallel arms.

The study is conducted as follows: eligible subjects are randomized parallelly into 3 arms. Each arm comprises 40 subjects orally receive active (FB-1603 165 mg oral capsule) or placebo (placebo capsule) two weeks before and eight weeks after TACE. Each subject will begin receiving FB-1603 oral capsule or placebo two weeks before TACE. As the appearance of the placebo capsule is identical to the FB-1603 165 mg oral capsule, study blinding will be maintained during the administration procedure. Other than staff involved in randomization, the sponsor, participants, and staff involved in the preparation of the study drug are blinded. Each subject is assigned to either active (FB-1603 165 mg oral capsule) or placebo treatment using a block randomization algorithm. Three times a day (TID) doses of FB-1603 165 mg oral capsule are escalated capsule low dose (990 mg/day) and high dose (1980 mg/day).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years (inclusive) of either gender
2. Willing and able to provide signed informed consent
3. Confirmed diagnosis of hepatocellular carcinoma by radiology, histology, or cytology
4. Subject has the willingness to undergo TACE
5. ECOG performance Status of 0-1
6. The patient is expected to survive more than 3 months
7. Laboratory values should meet all the following standards at the screening visit:

   A. AST, ALP and ALT are ≤ 5x ULN. B. International Normalized Ratio (INR) ≤ 1.5 C. Prothrombin time < 4 sec above upper limit of normal D. Absolute neutrophil count ≥ 1.5×10^9/L; Hemoglobin ≥ 9 g/dL; platelet ≥ 50×10^9/L.

   E. Total bilirubin < 2.5 mg/dL F. Serum creatinine < 2 mg/dL
8. With liver stiffness measurement >7 kPa (assessed by FibroScan®) or > 1.5 m/sec (assessed by acoustic radiation force impulse elastography (ARFI))

Exclusion Criteria:

1. Patients with evidence of macrovascular invasion
2. Patients with evidence of extrahepatic spread
3. Any condition representing a contraindication to TACE as determined by the investigators
4. Acute liver failure or liver function decompensation patient perform, such as hepatic encephalopathy, and ascites
5. Patients with acute or chronic active hepatitis B or C infection and are recommended to receive HBV or HCV treatment, e.g., Patient with HBV DNA ≥ 20,000 IU/ml or with detectable HCV RNA
6. Patients who have severe organic diseases on heart, lungs, brain, kidney, and gastrointestinal tract by the judgment of investigators
7. Patients with chronic pancreatitis
8. Patients who are taking any prohibited drugs that might interfere the trial
9. Patients who are not able to express the chief complaint, for example, the patients with psychosis and severe neurosis
10. Patients with active infections (infection requiring the use systemic antibiotics) within 4 weeks prior to the screening visit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2027-06-07 (Estimated); Study Completion 2027-08-06 (Estimated)

PRIMARY OUTCOMES:
Changes in the level of liver function | from baseline (day 0) to Visit 3 (day 4), Visit 4(day 7), Visit 5(day 10), and Visit 6(day 14)
  Changes in the level of liver function parameters, including aspartate transferase (AST), alanine transferase (ALT), or total bilirubin,

SECONDARY OUTCOMES:
Changes in the level of liver function | from baseline (day 0) to Visit 7 (day 28) and Visit 8 (day 56)
  Changes in the level of liver function parameters, including AST, ALT, or total bilirubin after TACE
Frequency and severity of adverse event (AE) during the study | up to 84 days
  Assessment of frequency and severity of adverse event (AE) during the study
Clinically significant changes in blood chemistry | from baseline (day 0) to Visit 3 (day 4), Visit 4 (day 7), Visit 5 (day 10), Visit 6 (day 14), Visit 7 (day 28), Visit 8 (day 56) and follow-up visit (day 84)
  Clinically significant changes in blood chemistry at each applicable visit
Clinically significant changes in coagulation test | from baseline (day 0) to Visit 3 (day 4), Visit 4 (day 7), Visit 5 (day 10), Visit 6 (day 14), Visit 7 (day 28), Visit 8 (day 56) and follow-up visit (day 84)
  Clinically significant changes in coagulation test at each applicable visit including international normalized ratio (INR) and prothrombin time.
Changes in measurements of indocyanine green retention (ICG) | from baseline (day 0) to Visit 3 (day 4) and Visit 5 (day 10)
  Changes in measurements of indocyanine green retention (ICG) test at each applicable visit
Level of liver fibrosis | at the screening visit (day -28 to -15), Visit 8 (day 56) and FV/ET (day 84)
  Level of liver fibrosis by elastography and fibrosis-4 (FIB-4) index
Incidence of postembolization syndrome | from baseline (day 0) to Visit 3 (day 4), Visit 4 (day 7), Visit 5 (day 10), Visit 6 (day 14), Visit 7 (day 28) and Visit 8 (day 56)
  Incidence of postembolization syndrome
Length of hospital stay after TACE | Visit 2 (day 0)
  Length of hospital stay after TACE
Changes in the level of quantitative HBsAg or HCV RNA | from screening visit (day -28 to -15) to Visit 8 (day 56) and FV/ET (day 84)
  Changes in the level of quantitative HBsAg or HCV RNA measured by PCR

CONTACTS AND LOCATIONS:
Overall Officials: Kai-Wen Huang, MD, MS, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan